CLINICAL TRIAL: NCT01375543
Title: Next Generation Sequencing to Identify Genetic Causes of Disease in Patients Participating in NICHD Clinical Protocols
Brief Title: Next Generation to Identify Genetic Causes of Disease in Patients Participating in NICHD Clinical Protocols
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110179; 11-CH-0179
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Genetic Predisposition
Keywords: Whole Exome; Whole Genome; Rare Disorders; Genetic Disorders
MeSH Terms: conditions — Genetic Predisposition to Disease; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Enrollees: Enrolled study participants in whom genetic sequencing was done

SUMMARY:
Background:

- The purpose of this study is to identify changes in genes that cause human diseases. We would like to obtain some of you or your child s DNA and test for changes in genes that may contribute to a disease in you or your family.

Objective:

-To allow for exomic or genomic sequencing of NICHD patients or family members in order to identify changes in genes that cause or contribute to a specific disease.

Eligibility:

* Children who are enrolled in an NICHD clinical study where the condition being studied may have a genetic cause.
* Family members of a child who is eligible for this study.

Design:

* Children and family members will supply DNA samples. If the samples are already available, no further DNA will be needed.
* If DNA is not available, samples of either blood or skin will be taken.
* We will use these samples with new DNA sequencing technology that looks at all the human genes we know about. This is known as exome and genome sequencing.

DETAILED DESCRIPTION:
Over the last few years advancements in DNA sequencing technology have progressed significantly. It now is feasible and economical to sequence the exome (known genes) or the entire genome. This technological advance can be applied to identifying genetic causes of rare diseases where traditional methods such as mapping frequently failed due to insufficient number of cases. These cases often present themselves in the context of other NICHD research protocols, such as teaching protocols, where it would not be efficient for the individual investigators to write a new protocol. It will also serve to standardize the consent document across NICHD for investigators that do not include exomic/genomic sequencing in their own protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Proband s that are enrolled in an NICHD clinical protocol for which there is a suspicion of an underlying genetic cause for a disease for which they are being evaluated.
  2. Family members of a proband who is eligible for this protocol.

EXCLUSION CRITERIA:

1. Normal volunteers unrelated to a proband with the disease of interest.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -Children who are enrolled in an NICHD clinical study where the condition being studied may have a genetic cause.@@@-Family members of a child who is eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2011-06-16 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Gene Mutations | Baseline, Continuously
  Identify genetic causes of rare diseases

SECONDARY OUTCOMES:
Deidentified sequence data | Baseline, Continuously
  Allow NICHD investigators to access de-identified sequence data generated by the NICHD Molecular Genomics Laboratory

CONTACTS AND LOCATIONS:
Overall Officials: An N Dang Do, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-CH-0179.html